CLINICAL TRIAL: NCT05161533
Title: CASPIAN-RT Trial: Hypofractionated Consolidative Radiation Therapy After Durvalumab (MEDI4736) Plus Platinum-Based Chemotherapy in Extensive Stage Small Cell Lung Cancer
Brief Title: Hypofractionated Radiation Therapy After Durvalumab and Chemotherapy for the Treatment of Stage IV Extensive Stage Small Cell Lung Cancer, CASPIAN-RT Trial
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed per SRC Low Accrual Policy. Study closed prior to any participants enrolled.
Sponsor: University of Washington (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1121732; NCI-2021-12429 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10810 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2021-12-01; First posted 2021-12-17 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-04

CONDITIONS: Extensive Stage Lung Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; durvalumab; Immunoglobulin G; Disulfides; Etoposide; Radiation Dose Hypofractionation; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (durvalumab, chemotherapy, radiation therapy) (Experimental): INDUCTION: Patients receive standard of care chemotherapy consisting of carboplatin or cisplatin and etoposide. Patients also receive durvalumab IV on day 1 of each cycle. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive durvalumab IV on day 1 of each cycle. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Beginning cycle 5 or 6 of durvalumab, patients undergo hypofractionated radiation therapy.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Biological: Durvalumab; Drug: Etoposide; Radiation: Hypofractionated Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated; Hypofractionated Radiotherapy; hypofractionation; Radiation, Hypofractionated
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well hypofractionated radiation therapy after durvalumab and chemotherapy works to shrink tumors in patients with stage IV extensive stage small cell lung cancer. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects than a conventionally fractionated radiation course. Immunotherapy with monoclonal antibodies, such as durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as carboplatin, cisplatin, and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Adding radiation after chemo and immunotherapy may help improve cancer control.

DETAILED DESCRIPTION:
OUTLINE:

INDUCTION: Patients receive standard of care chemotherapy consisting of carboplatin or cisplatin and etoposide. Patients also receive durvalumab intravenously (IV) on day 1 of each cycle. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive durvalumab IV on day 1 of each cycle. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Beginning cycle 5 or 6 of durvalumab, patients undergo hypofractionated radiation therapy.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >= 18 years at the time of screening
* Able to provide written informed which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol
* Histologically or cytologically documented extensive stage-small cell lung cancer (ES-SCLC) (American Joint Committee on Cancer [AJCC] 8th edition stage IV or tumor/nodal volume that is too large to be encompassed in a tolerable radiation plan). Staging scans must include brain imaging with a computed tomography (CT) w/ contrast or magnetic resonance imaging (MRI) head and body imaging with a CT chest/abdomen/pelvis or a positron emission tomography (PET)/CT
* Patients with brain metastases are eligible provided they are asymptomatic, or treated and stable off steroids and anticonvulsants for at least 1 month before study entry
* Patients must be considered suitable to receive a platinum-based chemotherapy regimen as first-line treatment for ES-SCLC. Chemotherapy must contain either carboplatin or cisplatin in combination with etoposide
* Eastern Cooperative Oncology Group (ECOG) performance-status score of 0-1 at enrollment
* Life expectancy >= 12 weeks at enrollment
* Body weight > 30 kg
* No prior exposure to immune-mediated therapy including, but not limited to, other anti-cytotoxic T-lymphocyte-associated antigen-4, anti-programmed cell death-1, anti-programmed cell death ligand-1, and anti-programmed cell death ligand-2 antibodies, excluding therapeutic anticancer vaccines, NOT INCLUDING if patients are currently within the first 4 cycles of chemotherapy and durvalumab for THIS diagnosis of ES-SCLC within the past 4 months
* Hemoglobin >= 9.0 g/dL (within 3 prior months)
* Absolute neutrophil count >= 1.5 x 10^9/L (within 3 prior months)
* Platelet count >= 75 x 10^9/L (within 3 prior months)
* Serum bilirubin =< 1.5 x the upper limit of normal (ULN) (within 3 prior months). This will not apply to patients with confirmed Gilbert's syndrome, who will be allowed in consultation with their physician
* In patients without hepatic metastasis: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN; for patients with hepatic metastases, ALT and AST =< 5 x ULN (within 3 prior months)
* Measured or calculated creatinine clearance: of > 40 mL/min as determined by Cockcroft-Gault (using actual body weight) (within 3 prior months)
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrhoeic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
  * Women >= 50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy)

Exclusion Criteria:

* Medical contraindication to platinum-etoposide
* Any anti-cancer therapies including chemotherapy, hormone therapy, or other immunotherapies in the 4 months prior to this diagnosis of ES-SCLC
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Any history of radiotherapy to the chest
* History of allogenic organ transplantation
* Has a peripheral nervous system (PNS) of autoimmune nature, requiring systemic treatment (systemic steroids or immunosuppressive agents) or has a clinical symptomatology suggesting worsening of PNS
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis with the exception of diverticulosis, systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome (granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, and uveitis, etc.). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, interstitial lung disease, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events or compromise the ability of the patient to give written informed consent
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease >= 5 years before the first dose of the investigational product and of low potential risk for recurrence
  * Adequately treated nonmelanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease (eg, cervical cancer in situ)
* History of leptomeningeal carcinomatosis
* History of active primary immunodeficiency
* Active infection, including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B virus (HBV) (known positive HBV surface antigen result), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of HBV core antibody and absence of HBV surface antigen) are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication). Premedication with steroids for chemotherapy is acceptable
* Receipt of live, attenuated vaccine within 30 days prior to the first dose of durvalumab. Patients, if enrolled, should not receive live vaccine whilst receiving durvalumab and up to 30 days after the last dose of durvalumab
* Female patients who are pregnant or breast-feeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-19 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Up to 3 years
  The distribution of time to event outcomes will be evaluated using the method of Kaplan-Meier. Confidence intervals for median times will be determined using the Brookmeyer-Crowley method. Confidence intervals around landmark times will be determined using Greenwood's formula for the variance and based on a log-log transformation applied on the survival function. Binary proportions will be calculated with associated confidence intervals for binary outcomes, such as response. Means and/or medians will be calculated for continuous outcomes. Confidence bounds will be provided for means and quartiles and ranges for median values. All confidence bounds will be presented as 95% bounds.

SECONDARY OUTCOMES:
Incidence of grade 2 or higher pneumonitis | Up to 90 days after the last dose of durvalumab
  The incidence of grade 2 or worse pneumonitis attributable to treatment will be evaluated and compared against the CASPIAN trial results. All toxicities of all grades will be monitored on study and reported. Binary proportions will be calculated with associated confidence intervals for binary outcomes, such as toxicity.
Overall survival | Up to 3 years
  The distribution of time to event outcomes will be evaluated using the method of Kaplan-Meier. Confidence intervals for median times will be determined using the Brookmeyer-Crowley method. Confidence intervals around landmark times will be determined using Greenwood's formula for the variance and based on a log-log transformation applied on the survival function. Binary proportions will be calculated with associated confidence intervals for binary outcomes, such as response. Means and/or medians will be calculated for continuous outcomes. Confidence bounds will be provided for means and quartiles and ranges for median values. All confidence bounds will be presented as 95% bounds.
Response rate | Up to 3 years
  The distribution of time to event outcomes will be evaluated using the method of Kaplan-Meier. Confidence intervals for median times will be determined using the Brookmeyer-Crowley method. Confidence intervals around landmark times will be determined using Greenwood's formula for the variance and based on a log-log transformation applied on the survival function. Binary proportions will be calculated with associated confidence intervals for binary outcomes, such as response. Means and/or medians will be calculated for continuous outcomes. Confidence bounds will be provided for means and quartiles and ranges for median values. All confidence bounds will be presented as 95% bounds.
Healthcare related quality of life: EORTC QLQ-C30 | Up to 3 years
  Will be measured by European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30).
Healthcare related quality of life: EORTC QLQ-LC13 | Up to 3 years
  Will be measured by European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire - QLQ-Lung Cancer (LC)13 (EORTC QLQ-LC13).

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zeng, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No